CLINICAL TRIAL: NCT00516620
Title: Fruits, Vegetables, and Whole Grains: A Community-based Intervention
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Unity Health Toronto (Other); Cancer Care Ontario (Other)
Responsible Party: Principal Investigator, David Jenkins, Professor, University of Toronto
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: REB 04-016C; CIHR-NET 105919
Record Dates: First submitted 2007-08-13; First posted 2007-08-15 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Heart Disease; Diabetes; Hypertension
Keywords: Body Weight
MeSH Terms: conditions — Heart Diseases; Diabetes Mellitus; Hypertension; Body Weight | interventions — Fruit; Vegetables; Whole Grains; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Participants receive Health Canada's Food Guide and Physical Activity guide.
  Interventions: Behavioral: No further instruction; Behavioral: Food Delivery; Behavioral: Fruits (F), vegetables (V), and whole grain (WG) counseling; Behavioral: Counseling to reduce soft drink intake.; Behavioral: Food Delivery & F, V & WG counseling.; Behavioral: Food delivery & soft drink counseling; Behavioral: F, V, WG & soft drink counseling; Behavioral: Food delivery and F,V, WG & soft drink counseling
- 2 (Active Comparator): Participants receive a weekly sample food basket for 6 months consisting of fruits, vegetables, whole grains, and vegetable protein products.
  Interventions: Behavioral: Food Delivery; Behavioral: Food Delivery & F, V & WG counseling.; Behavioral: Food delivery & soft drink counseling; Behavioral: Food delivery and F,V, WG & soft drink counseling
- 3 (Active Comparator): Participants receive intensive dietary counseling for 6 months to increase intake of fruits, vegetables, whole grains, and vegetable protein products.
  Interventions: Behavioral: Fruits (F), vegetables (V), and whole grain (WG) counseling; Behavioral: Food Delivery & F, V & WG counseling.; Behavioral: F, V, WG & soft drink counseling; Behavioral: Food delivery and F,V, WG & soft drink counseling
- 4 (Active Comparator): Participants receive intensive dietary counseling for 6 months to decrease intake of sweetened soft drink.
  Interventions: Behavioral: Counseling to reduce soft drink intake.; Behavioral: Food delivery & soft drink counseling; Behavioral: F, V, WG & soft drink counseling; Behavioral: Food delivery and F,V, WG & soft drink counseling

INTERVENTIONS:
Behavioral: No further instruction — Participants receive Health Canada's Food Guide and Physical Activity Guide and no other intervention for the 6 months of the intervention period.
  Other Names: Control
  Arms: 1
Behavioral: Food Delivery — Participants receive Canada's Food Guide and Physical Activity guide, in addition to a a weekly sample food basket for 6 months consisting of fruits, vegetables, whole grains, and vegetable protein products.
  Arms: 1; 2
Behavioral: Fruits (F), vegetables (V), and whole grain (WG) counseling — Participants receive Canada's Food Guide and Physical Activity guide, and intensive dietary counseling for 6 months to increase intake of fruits, vegetables, whole grains, and vegetable protein products. The counselling frequency will be weekly intervals for the first month, and then monthly sessions for the second to sixth months.
  Other Names: Fruit, Vegetable and Whole Grain Counseling
  Arms: 1; 3
Behavioral: Counseling to reduce soft drink intake. — Participants receive Health Canada's Food Guide and Physical Activity guide, and intensive dietary counseling for 6 months to decrease intake of sweetened soft drink. The counselling frequency will be weekly intervals for the first month, and then monthly sessions for the second to sixth months.
  Other Names: Sweetened Soft Drink Counseling
  Arms: 1; 4
Behavioral: Food Delivery & F, V & WG counseling. — Participants receive Health Canada's Food Guide and Physical Activity guide, a weekly sample food basket for 6 months consisting of fruits, vegetables, whole grains, and vegetable protein products, and intensive dietary counseling to increase intake of fruits, vegetables, whole grains, and vegetable protein products. The counselling frequency will be weekly intervals for the first month, and then monthly sessions for the second to sixth months.
  Other Names: Food Delivery, Fruit, Vegetable and Whole Grain Counseling
  Arms: 1; 2; 3
Behavioral: Food delivery & soft drink counseling — Participants receive Health Canada's Food Guide and Physical Activity guide, a weekly sample food basket for 6 months consisting of fruits, vegetables, whole grains, and vegetable protein products, and intensive dietary counseling for 6 months to decrease intake of sweetened soft drink. The counselling frequency will be weekly intervals for the first month, and then monthly sessions for the second to sixth months.
  Other Names: Food Delivery, and Sweetened Soft Drink Counseling
  Arms: 1; 2; 4
Behavioral: F, V, WG & soft drink counseling — Participants receive Health Canada's Food Guide and Physical Activity guide, and intensive dietary counseling for 6 months to increase intake of fruits, vegetables, whole grains, and vegetable protein products, and also to decrease intake of sweetened soft drink. The counseling frequency will be weekly intervals for the first month, and then monthly sessions for the second to sixth months.
  Other Names: Fruit, Vegetable, Whole Grain, Sweetened Soft Drink Counseling
  Arms: 1; 3; 4
Behavioral: Food delivery and F,V, WG & soft drink counseling — Participants receive Health Canada's Food Guide and Physical Activity guide, receive a weekly sample food basket for 6 months consisting of fruits, vegetables, whole grains, and vegetable protein products, and intensive dietary counseling for 6 months to increase intake of fruits, vegetables, whole grains, and vegetable protein products, and also to decrease intake of sweetened soft drink. The counselling frequency will be weekly intervals for the first month, and then monthly sessions for the second to sixth months.
  Other Names: Food Delivery, Fruit, Vegetable, Whole Grain, and Sweetened Soft Drink Counseling

SUMMARY:
The aim of this study is to see if the investigators can encourage people to eat more fruits, vegetables and whole grains and drink less pop by giving them advice about their diet, or by providing them with samples of different kinds of foods. The investigators are interested in the effect this has on reducing the risk of chronic disease. The investigators will also be investigating how certain genes affect the choices people make about the foods they eat.

DETAILED DESCRIPTION:
Governments and major national agencies throughout the western world concerned with chronic disease prevention (heart disease, stroke, diabetes, and cancer) uniformly advocate increased intakes of fruit, vegetables and whole grain cereals. All also agree that body weight reduction is central to reducing the risk of heart disease, stroke, type 2 diabetes, and certain cancers. Nevertheless, there is no official advice encouraging increased consumption of these foods in order to achieve and maintain a healthy body weight. Most importantly, there are no intervention studies that have tested the assumption that increased intake of fruit, vegetables and whole grain cereals will promote a healthier body weight. Our study will therefore address this issue to determine the effect of an increased intake of fruit, vegetables, and whole grain cereals on body weight, the intensity of effort required to achieve compliance, the durability of this habit, genetic determinants, and the effect on biomarkers of chronic disease risk.

We will ask approximately 780 families to take part in this study. We will invite households to take part if there is at least one adult who is eligible for our study, and who agrees to participate.

To be eligible for this study, participants must be at least 18 years old and have no medical conditions that would make it unsafe for them to take part. Before beginning the study, the medical history and other measures will be checked to ensure participant safety and suitability for participating in the study.

This study consists of three parts. If agreement to participate is given, the first part is to make an appointment to come to our study clinic to give a fasting blood sample (baseline measurements), about 40mL of blood. The clinic visit will last approximately 40 minutes. All participants will be asked to complete a short checklist about their medical history, which includes information to make sure that they and their household are eligible for participation. Body fat measurements will also be made using a non-invasive, very simple machine called Futrex as well as height, weight, waist-to-hip ratio, and blood pressure. Part of the blood sample will be used for a health screen to ensure subject safety and suitability for participating in the study. Blood samples will be stored in a secured location and analyzed at the end of the study for cholesterol levels and other risk factors for heart disease. Part of the blood sample will be used in DNA analysis to help us understand the genes related to food intake and metabolism. We will also ask all participants to complete a questionnaire package about their eating habits and their physical activity either prior to the clinic visit or at the end of the clinic visit. Once the questionnaires are completed and returned to the study office, the second part of the study will commence.

The second part is the intervention itself, lasting six months. If households are deemed to be eligible, they will be 'randomized' into one of eight study groups with all groups receiving Canada's Food Guide & Physical Activity Guide. The study groups involve a combination of different kinds of dietary advice and provision of fruit, vegetables, and whole grain cereals.

* Treatment 1: no food provision or dietary advice.
* Treatment 2: food delivery.
* Treatment 3: counseling on fruit, vegetables and whole grains.
* Treatment 4: counseling to reduce soft drink intake.
* Treatment 5: food delivery AND counseling on fruit, vegetables and whole grains.
* Treatment 6: food delivery AND counseling to reduce soft drink intake.
* Treatment 7: counseling on fruit, vegetables, whole grains AND counseling on the reduction of soft drink intake.
* Treatment 8: food delivery AND counseling on fruit, vegetables, whole grains AND counseling on the reduction of soft drink intake.

All food boxes are prepared and delivered by Food Share, a Toronto-based non-profit organization that has an existing system for home delivery of nutritious food boxes. If participants do receive dietary counseling, it will involve a phone call once a week for the first month (for about 20 minutes) then a phone call once a month for the next 5 months. At the end of six months, participants will be asked to fill in provided questionnaires and return to the clinic to repeat the procedures.

The third part is a follow-up 12 months after the end of the intervention. Again, participants will be asked to fill in provided questionnaires and return to the clinic to repeat the procedures.

ELIGIBILITY:
Inclusion Criteria:

* residents of households within the City of Toronto 416 calling area
* respond to advertisements in newspaper, on radio, and from flyers
* Eligible households will include at least one willing adult 18 years or older; able to communicate in English, at least one adult with BMI >/= 25
* Pregnant and breastfeeding mothers who fit the criteria above are eligible to join the study 6 months post-partum or 6 months after the cessation of breastfeeding
* Individuals who fit the inclusion criteria but recently (past 6 months) started blood pressure medication are eligible for the study once their blood pressure is under control
* Individuals who fit the inclusion criteria but recently started hypothyroid medication or diuretics will be eligible after 1 month of treatment

Exclusion Criteria:

* Residing outside of the 416 area code
* under 18 years of age
* actively following a special diet or weight-loss program
* major cardiovascular event in the previous 6 months
* recently (past 6 months) started blood pressure medication
* diabetes, liver disease, renal failure, cancer (or a history of malignancy), inflammatory bowel disease, individuals with acute or chronic infections, either bacterial or viral, or individuals suffering from chronic inflammatory diseases, irritable bowel syndrome, peanut or nut allergy, major surgery in the previous 6 months
* blood pressure greater than 145/95 on repeated measurements will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 960 (Actual)
Dates: Start 2005-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Body Weight | 18 months

SECONDARY OUTCOMES:
Biomarkers of diet and obesity-related chronic diseases (serum lipids, homocysteine and C-reactive protein) and genotypes | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Daivd JA Jenkins, MD, PhD, Principal Investigator — University of Toronto, St. Michael's Hospital
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Jamnik J, Villa CR, Dhir SB, Jenkins DJA, El-Sohemy A. Prevalence of positive coeliac disease serology and HLA risk genotypes in a multiethnic population of adults in Canada: a cross-sectional study. BMJ Open. 2017 Oct 6;7(10):e017678. doi: 10.1136/bmjopen-2017-017678. PMID 39272232
- [Derived] Wang J, Jamnik J, Garcia-Bailo B, Nielsen DE, Jenkins DJA, El-Sohemy A. ABO Genotype Does Not Modify the Association between the "Blood-Type" Diet and Biomarkers of Cardiometabolic Disease in Overweight Adults. J Nutr. 2018 Apr 1;148(4):518-525. doi: 10.1093/jn/nxx074. PMID 29659952
- [Derived] Jenkins DJA, Boucher BA, Ashbury FD, Sloan M, Brown P, El-Sohemy A, Hanley AJ, Willett W, Paquette M, de Souza RJ, Ireland C, Kwan N, Jenkins A, Pichika SC, Kreiger N. Effect of Current Dietary Recommendations on Weight Loss and Cardiovascular Risk Factors. J Am Coll Cardiol. 2017 Mar 7;69(9):1103-1112. doi: 10.1016/j.jacc.2016.10.089. PMID 28254171